CLINICAL TRIAL: NCT00962845
Title: A Phase 0 Trial of Hydroxychloroquine, an Inhibitor of Autophagy, in Patients With Stage III or IV Resectable Melanoma
Brief Title: Hydroxychloroquine in Patients With Stage III or Stage IV Melanoma That Can Be Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0220090117; P30CA072720 (NIH); CDR0000648156 (Other: NIH); NCI-2011-03324 (Other: CTRP (Clinical Trials Reporting System)); 090901 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxychloroquine (Experimental): Patients must have tumor accessible for pre-treatment biopsy (see 5.1.2). Patients will be enrolled on the trial, undergo biopsy of their tumors if no banked tumor is available, and then begin an oral dose of HCQ at the dose of 200 mg twice daily. At the end of two weeks the patients will undergo resection of their tumors. HCQ will be given to the patients up to the day of the operation but not resumed postoperatively.
  Interventions: Drug: hydroxychloroquine

INTERVENTIONS:
Drug: hydroxychloroquine — 200 mg twice daily in the first ten patients. If the first ten patients tolerate this dosage schedule (200 mg bid) without significant side effects (Grade 3 or greater gastrointestinal upset, skin toxicity, myopathy or any visual disturbances whatsoever), the second ten patients will be enrolled at a dose of 400 mg bid

SUMMARY:
RATIONALE: Studying samples of blood, tumor tissue, and skin in the laboratory from patients with melanoma receiving hydroxychloroquine may help doctors understand the effect of hydroxychloroquine on biomarkers.

PURPOSE: This early phase I trial is studying hydroxychloroquine in patients with stage III or stage IV melanoma that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To characterize the effects of hydroxychloroquine (HCQ) on the modulation of markers of autophagy, as measured by p62, Beclin1, LC3, and GRp170 expression, in pre- and post-treatment tumor biopsy samples, skin samples, and peripheral blood mononuclear cell samples from patients with stage III or IV melanoma undergoing palliative or curative surgery.

Secondary

* To determine whether the steady-state plasma concentration of HCQ correlates with observed trends in induced markers of autophagy.
* To determine the potential mechanisms of antitumor effect of HCQ, as measured by a reduction in tumor cell proliferation (Ki-67 and mitotic rate) or an increase in apoptosis (activated caspase-3 and TUNEL assays) in melanoma specimens.

OUTLINE: Patients receive oral hydroxychloroquine twice daily for 14 days in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

Blood, tumor tissue, and skin samples are collected for pharmacokinetic and correlative laboratory studies. Expression of p62, Beclin1, LC3, and GRp170 (autophagy markers) is analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed melanoma

  * Stage III or IV disease
  * Has ≥ 2 resectable tumors OR tumor large enough to undergo pre-treatment core needle biopsy
* Must be a candidate for curative or palliative surgical resection of disease
* Brain metastases allowed provided they were previously treated and have been stable for > 2 weeks

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count > 1,500/mm³
* Platelet count > 100,000/mm³
* SGOT and SGPT < 2.5 times upper limit of normal (ULN)
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of any social or medical condition that, in the opinion of the investigator, may interfere with the patient's ability to comply with the study or pose additional or unacceptable risk to the patient
* No concurrent serious systemic disorder that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to complete the study
* No active clinically significant infection requiring antibiotics
* No hypertension that cannot be controlled by medication (i.e., diastolic blood pressure > 100 mm Hg despite optimal medical therapy)
* No pre-existing thyroid abnormality with thyroid-stimulating hormone that cannot be maintained in the normal range with medication
* No known HIV positivity
* No psoriasis or porphyria
* No known hypersensitivity to 4-aminoquinoline compounds
* No retinal or visual field changes from prior 4-aminoquinoline compound use
* No known G-6P deficiency
* No known gastrointestinal pathology that would interfere with drug bioavailability
* No known prior hypersensitivity to hydroxychloroquine or any of its components
* No clinically significant bleeding or clotting disorder that would preclude curative or palliative surgery

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 2 weeks since prior cytotoxic or biologic agents (6 weeks for mitomycin or nitrosoureas)
* At least 2 weeks since prior surgery, radiotherapy, hormonal therapy, or other drug therapy for melanoma
* No concurrent treatment for rheumatoid arthritis or systemic lupus erythematosus
* No concurrent disease-modifying anti-rheumatic drugs
* No concurrent hydroxychloroquine for treatment or prophylaxis of malaria
* No concurrent aurothioglucose or antimalarial agents
* No other concurrent chemotherapy, immunotherapy, hormonal therapy, radiotherapy, or surgery for cancer
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05-30 (Actual); Study Completion 2013-05-30 (Actual)

PRIMARY OUTCOMES:
Modulation of markers of autophagy by hydroxychloroquine (HCQ), as measured by p62, Beclin1, LC3, and GRp170 expression | 1 year

SECONDARY OUTCOMES:
Correlation of steady-state plasma concentration of HCQ with observed trends in induced markers of autophagy | 1 year
Potential mechanisms of antitumor effect of HCQ, as measured by a reduction in tumor cell proliferation or an increase in apoptosis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Janice M. Mehnert, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States